CLINICAL TRIAL: NCT04046055
Title: Cerebellar Transcranial Direct Current Stimulation in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thorsten Rudroff (Other)
Responsible Party: Sponsor-Investigator, Thorsten Rudroff, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201906759
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease; Brain Stimulation; Cerebellum
Keywords: transcranial direct current stimulation; walking; balance
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All participants completed all 5 randomly ordered tDCS sessions (sham, unilateral 2 mA, unilateral4 mA, bilateral 2 mA, and bilateral 4 mA.
Masking Description: Participants will be blind to the different stimulation intensities (sham, 2 mA, 4 mA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sham and Experimental Sessions (Experimental): 50% of participants will have a unilateral cerebellar montage with the anode (active electrode) three cm lateral to the inion on the side ipsilateral to the more PD-affected side and the cathode (return electrode) on the ipsilateral cheek. 50% of participants will have a bilateral cerebellar tDCS will have both electrodes placed 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is turned (2 mA) on for the 30 seconds at the beginning and the end of the trial, but it turned to 0 mA in the intervening time.
  A unilateral cerebellar montage will be applied. tDCS intensity will be 2 mA. Bilateral cerebellar tDCS will be applied. tDCS intensity will be 2 mA. A unilateral cerebellar montage will be applied. tDCS intensity will be 4 mA. Bilateral cerebellar tDCS will be applied. tDCS intensity will be 4 mA.
  Interventions: Device: Transcranial direct current stimulation at 2 mA; Device: Transcranial direct current stimulation at 4 mA; Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation at 2 mA — Uses weak electrical current (2 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
  Other Names: tDCS
Device: Transcranial direct current stimulation at 4 mA — Uses weak electrical current (4 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
  Other Names: tDCS
Device: Sham transcranial direct current stimulation — Uses weak electrical current (2 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo-like effects or participant expectation bias.
  Other Names: Sham tDCS

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder and affects approximately 1 million people in the United States with total annual costs approaching 11 billion dollars. The most common symptoms of PD are tremor, stiffness, slowness, and trouble with balance/walking, which lead to severe impairments in performing activities of daily living. Current medical and surgical treatments for PD are either only mildly effective, expensive, or associated with a variety of side-effects. Therefore, the development of practical and effective add-ons to current therapeutic treatment approaches would have many benefits. Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that can affect brain activity and can help make long-term brain changes to improve functions like walking and balance. While a few initial research studies and review articles involving tDCS have concluded that tDCS may improve PD walking and balance, many results are not meaningful in real life and several crucial issues still prevent tDCS from being a useful add-on intervention in PD. These include the selection of stimulation sites (brain regions stimulated) and tDCS electrode placement. Most studies have targeted the motor cortex (brain region that controls intentional movement), but there is evidence that the cerebellum - which helps control gait and balance, is connected to several other brain areas, and is easily stimulated with tDCS - may be a likely location to further optimize walking and balance in PD. There is also evidence that certain electrodes placements may be better than others. Thus, the purpose of this study is to determine the effects of cerebellar tDCS stimulation using two different placement strategies on walking and balance in PD.

Additionally, although many tDCS devices are capable of a range of stimulation intensities (for example, 0 mA - 5 mA), the intensities currently used in most tDCS research are less than 2 mA, which is sufficient to produce measurable improvements; but, these improvements may be expanded at higher intensities. In the beginning, when the safety of tDCS was still being established for human subjects, careful and moderate stimulation approaches were warranted. However, recent work using stimulation at higher intensities (for example, up to 4 mA) have been performed in different people and were found to have no additional negative side-effects. Now that the safety of tDCS at higher intensities is better established, studies exploring the differences in performance between moderate (i.e., 2 mA) and higher (i.e., 4 mA) intensities are necessary to determine if increasing the intensity increases the effectiveness of the desired outcome.

Prospective participants will include 10 people with mild-moderate PD that will be recruited to complete five randomly-ordered stimulation sessions, separated by at least 5 days each. Each session will involve one visit to the Integrative Neurophysiology Laboratory (INPL) and will last for approximately one hour. Data collection is expected to take 4-6 months. Each session will include walking and balance testing performed while wearing the tDCS device. Total tDCS stimulation time for each session will be 25 minutes.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder and affects approximately 1 million people in the United States with total annual costs approaching 11 billion dollars. The most common symptoms of PD are tremor, stiffness, slowness, and trouble with balance/walking, which lead to severe impairments in performing activities of daily living. Current medical and surgical treatments for PD are either only mildly effective, expensive, or associated with a variety of side-effects. Therefore, the development of practical and effective add-ons to current therapeutic treatment approaches would have many benefits. Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that can affect brain activity and can help make long-term brain changes to improve functions like walking and balance. While a few initial research studies and review articles involving tDCS have concluded that tDCS may improve PD walking and balance, many results are not meaningful in real life and several crucial issues still prevent tDCS from being a useful add-on intervention in PD. These include the selection of stimulation sites (brain regions stimulated) and tDCS electrode placement. Most studies have targeted the motor cortex (brain region that controls intentional movement), but there is evidence that the cerebellum - which helps control gait and balance, is connected to several other brain areas, and is easily stimulated with tDCS - may be a likely location to further optimize walking and balance in PD. There is also evidence that certain electrodes placements may be better than others. Thus, the purpose of this study is to determine the effects of cerebellar tDCS stimulation using two different placement strategies on walking and balance in PD.

Additionally, although many tDCS devices are capable of a range of stimulation intensities (for example, 0 mA - 5 mA), the intensities currently used in most tDCS research are less than 2 mA, which is sufficient to produce measurable improvements; but, these improvements may be expanded at higher intensities. In the beginning, when the safety of tDCS was still being established for human subjects, careful and moderate stimulation approaches were warranted. However, recent work using stimulation at higher intensities (for example, up to 4 mA) have been performed in different people and were found to have no additional negative side-effects. Now that the safety of tDCS at higher intensities is better established, studies exploring the differences in performance between moderate (i.e., 2 mA) and higher (i.e., 4 mA) intensities are necessary to determine if increasing the intensity increases the effectiveness of the desired outcome.

Prospective participants will include 10 people with mild-moderate PD that will be recruited to complete five randomly-ordered stimulation sessions (baseline/SHAM, unilateral tDCS montage at 2 mA, unilateral tDCS montage at 4 mA, bilateral tDCS montage at 2 mA, and bilateral montage at 4 mA), separated by at least 5 days. Each session will involve one visit to the Integrative Neurophysiology Laboratory (INPL) and will last for approximately one hour. Data collection is expected to take 4-6 months. Each session will include gait (30-meter walk test [30mWT], 6-minute walk test [6MWT], Timed Up and Go [TUG]) and balance testing (standing on a force platform with either a firm surface or a foam surface) performed in conjunction with one of the five randomly-ordered stimulation conditions (SHAM, unilateral 2 mA, unilateral 4 mA, bilateral 2 mA, and bilateral 4 mA). Total tDCS stimulation time for each session will be 25 minutes. Gait characteristics (i.e., gait speed, stride length, step length, toe-off angle, etc.) and distance walked during the 30mWT and 6MWT will also be determined with inertial sensors (OPAL motion sensors).

ELIGIBILITY:
Inclusion Criteria:

* 1) Adult (50-90 yrs) with a positive diagnosis of Parkinson's disease from a movement disorder specialist
* 2) an unchanged regimen of dopaminergic medication for at least the last 3 months
* 3) able to independently walk for 6 min
* 4) without other chronic psychiatric or medical conditions
* 5) not taking any psychoactive medications

Exclusion Criteria:

* 1) pregnant
* 2) known holes or fissures in the skull
* 3) metallic objects or implanted devices in the skull (e.g., metal plate, deep brain stimulator)
* 4) current or previous injuries or surgeries that cause unusual gait
* 5) score less than 24 or 17 on the Montreal Cognitive Assessment or telephone-Montreal Cognitive Assessment, respectively
* 6) experience freezing of gait
* 7) a diagnosis of dementia or other neurodegenerative diseases

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Rudroff, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects in this study completed all of the study arms (repeated-measure design).
Groups:
- Sham/2mA/ Unilateral 2 mA/ Bilateral 2 mA/ Unilateral 4 mA /Bilateral 4 mA): Sham transcranial direct current stimulation: Uses weak electrical current (2 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo-like effects or participant expectation bias.
  A unilateral cerebellar montage with the anode three cm lateral to the inion on the side ipsilateral to the more PD-affected side and the cathode on the ipsilateral cheek. Stimulation is ramped up to 2 mA or 4 mA over the first 30 seconds and stays at 2 mA for the remainder of the stimulation time.
  Bilateral cerebellar tDCS will have both electrodes placed 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is ramped up to 2 mA over the first 30 seconds and stays at 2 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 2 mA/4mA: Uses weak electrical current to either increase or decrease brain excitability and improve functional or cognitive outcomes.
Period: Overall Study
Arm/Group | Sham/2mA/ Unilateral 2 mA/ Bilateral 2 mA/ Unilateral 4 mA /Bilateral 4 mA)
Started | 7
Sham | 7
Unilateral, 2 mA | 7
Bilateral, 2 mA | 7
Unilateral, 4 mA | 7
Bilateral, 4 mA | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham, Unilateral 2 mA, Bilateral 2 mA, Unilateral 4 mA, and Bilateral 4 mA): Sham transcranial direct current stimulation: Uses weak electrical current (2 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo-like effects or participant expectation bias.
  A unilateral cerebellar montage with the anode three cm lateral to the inion on the side ipsilateral to the more PD-affected side and the cathode on the ipsilateral cheek. Stimulation is ramped up to 2 mA over the first 30 seconds and stays at 2 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 2 mA/4mA: Uses weak electrical current to either increase or decrease brain excitability and improve functional or cognitive outcomes.
  Bilateral cerebellar tDCS will have both electrodes placed 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is ramped up to 2 mA over the first 30 seconds and stays at 2 mA/4mA for the remainder of the stimulation time.
Arm/Group | Sham, Unilateral 2 mA, Bilateral 2 mA, Unilateral 4 mA, and Bilateral 4 mA)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
UPDRS-III [Mean (Standard Deviation); unit: Scores on scale] — Scores range from zero (i.e., no motor symptoms) to 132 (i.e., severe motor symptoms. Lower mean values indicate that PD less-sever symptoms and higher mean values indicate more severe symptoms.
  There is no accepted "cut-off" value(s) to stratify symptom severity. In this study, such a value is even less relevant because we investigated how changes in these scores (i.e., within a given subject) changed from intervention to intervention. Thus, a lower relative score in one condition might indicate improved symptoms from that condition's intervention compared to those with higher scores.
  Scores on scale | 32.6 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Speed Walked During 30 Meter Walk Test
Description: Walk as fast and as safe as possible over 30 meter
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Groups:
- Sham 4 mA: Sham transcranial direct current stimulation: Uses weak electrical current (2 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo-like effects or participant expectation bias.
- Unilateral 2 mA: A unilateral cerebellar montage with the anode three cm lateral to the inion on the side ipsilateral to the more PD-affected side and the cathode on the ipsilateral cheek. Stimulation is ramped up to 2 mA over the first 30 seconds and stays at 2 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 2 mA: Uses weak electrical current to either increase or decrease brain excitability and improve functional or cognitive outcomes.
- Bilateral 2 mA: Bilateral cerebellar tDCS will have both electrodes placed 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is ramped up to 2 mA over the first 30 seconds and stays at 2 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 2 mA: Uses weak electrical current to either increase or decrease brain excitability and improve functional or cognitive outcomes.
- Unilateral 4 mA: A unilateral cerebellar montage with the anode three cm lateral to the inion on the side ipsilateral to the more PD-affected side and the cathode on the ipsilateral cheek. Stimulation is ramped up to 4 mA over the first 30 seconds and stays at 4 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 4 mA: Uses weak electrical current to either increase or decrease brain excitability and improve functional or cognitive outcomes.
- Bilateral 4 mA: Bilateral cerebellar tDCS will have both electrodes placed 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is ramped up to 4 mA over the first 30 seconds and stays at 4 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 4 mA: Uses weak electrical current to either increase or decrease brain excitability and improve functional or cognitive outcomes.
Arm/Group | Sham 4 mA | Unilateral 2 mA | Bilateral 2 mA | Unilateral 4 mA | Bilateral 4 mA
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
meters per second (m/s) | 5.63 (0.84) | 5.65 (1.04) | 5.77 (1.07) | 5.86 (1.06) | 5.77 (1.24)

2. Primary Outcome: Time to Complete the Timed Up and Go Test
Description: From a seated position, stand up, walk 5 meters, turn around, walk back, and sit back down in the chair.
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: seconds (s)
Groups:
- Sham: Sham transcranial direct current stimulation: Uses weak electrical current (2 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo-like effects or participant expectation bias.
Arm/Group | Sham | Unilateral 2 mA | Bilateral 2 mA | Unilateral 4 mA | Bilateral 4 mA
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
seconds (s) | 11.9 (2.7) | 12.43 (2.32) | 12.80 (2.42) | 12.42 (2.72) | 12.70 (3.28)

3. Primary Outcome: Movement of the Center of Pressure (2D; Forward-backward, Left-right) While Standing on a Firm Surface (Force Platform) for 1 Minute
Description: Stand as still as possible on a firm surface for 1 minute with the eyes open. Calculate the area of an ellipse that contains 95% of the 2D trace of the center of pressure movement.
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: centimeters squared (cm^2)
Arm/Group | Sham | Unilateral 2 mA | Bilateral 2 mA | Unilateral 4 mA | Bilateral 4 mA
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
centimeters squared (cm^2) | 3.22 (2.56) | 2.47 (2.34) | 1.72 (0.50) | 1.60 (0.74) | 1.57 (0.39)

4. Primary Outcome: Movement of the Center of Pressure (2D; Forward-backward, Left-right) While Standing on a Foam Surface (6 cm Foam Pad Placed on Top of Force Platform) for 1 Minute
Description: Stand as still as possible on a foam surface for 1 minute with the eyes open. Calculate the area of an ellipse that contains 95% of the 2D trace of the center of pressure movement.
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: centimeters squared (cm^2)
Arm/Group | Sham | Unilateral 2 mA | Bilateral 2 mA | Unilateral 4 mA | Bilateral 4 mA
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
centimeters squared (cm^2) | 8.34 (7.57) | 7.53 (4.35) | 9.36 (6.90) | 8.30 (6.40) | 7.60 (3.63)

5. Secondary Outcome: Movement of the Center of Pressure (1D; Forward-backward) While Standing on a Firm Surface (Force Platform) for 1 Minute
Description: Stand as still as possible on a firm surface for 1 minute with the eyes open.
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Sham | Unilateral 2 mA | Bilateral 2 mA | Unilateral 4 mA | Bilateral 4 mA
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
centimeters (cm) | 2.38 (0.70) | 2.90 (0.91) | 2.25 (0.62) | 2.25 (0.69) | 2.86 (1.02)

6. Secondary Outcome: Movement of the Center of Pressure (1D; Left-Right) While Standing on a Firm Surface (Force Platform) for 1 Minute
Description: Stand as still as possible on a firm surface for 1 minute with the eyes open.
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Sham | Unilateral 2 mA | Bilateral 2 mA | Unilateral 4 mA | Bilateral 4 mA
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
centimeters (cm) | 2.1 (1.8) | 1.4 (0.6) | 1.3 (0.3) | 1.1 (0.4) | 1.1 (0.4)

7. Secondary Outcome: Movement of the Center of Pressure (1D; Forward-backward) While Standing on a Foam Surface (6 cm Foam Pad Placed on Top of Force Platform) for 1 Minute
Description: Stand as still as possible on a foam surface for 1 minute with the eyes open.
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Sham | Unilateral 2 mA | Bilateral 2 mA | Unilateral 4 mA | Bilateral 4 mA
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
centimeters (cm) | 4.4 (2.8) | 4.0 (1.1) | 4.5 (1.8) | 4.11 (1.41) | 4.08 (1.19)

8. Secondary Outcome: Movement of the Center of Pressure (1D; Left-Right) While Standing on a Foam Surface (6 cm Foam Pad Placed on Top of Force Platform) for 1 Minute
Description: Stand as still as possible on a foam surface for 1 minute with the eyes open.
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Sham | Unilateral 2 mA | Bilateral 2 mA | Unilateral 4 mA | Bilateral 4 mA
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
centimeters (cm) | 3.6 (1.8) | 3.4 (1.0) | 3.3 (1.3) | 3.3 (1.2) | 3.3 (1.0)

ADVERSE EVENTS:
Time Frame: 5 weeks
Groups:
- Sham: 50% of participants will have a unilateral cerebellar montage with the anode (active electrode) three cm lateral to the inion on the side ipsilateral to the more PD-affected side and the cathode (return electrode) on the ipsilateral cheek. 50% of participants will have a bilateral cerebellar tDCS will have both electrodes placed 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is turned (2 mA) on for the 30 seconds at the beginning and the end of the trial, but it turned to 0 mA in the intervening time.
  Sham transcranial direct current stimulation: Uses weak electrical current (2 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo-like effects or participant expectation bias.
- Unilateral, 2 mA: A unilateral cerebellar montage with the anode three cm lateral to the inion on the side ipsilateral to the more PD-affected side and the cathode on the ipsilateral cheek. Stimulation is ramped up to 2 mA over the first 30 seconds and stays at 2 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 2 mA: Uses weak electrical current (2 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
- Bilateral, 2 mA: Bilateral cerebellar tDCS will have both electrodes placed 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is ramped up to 2 mA over the first 30 seconds and stays at 2 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 2 mA: Uses weak electrical current (2 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
- Unilateral, 4 mA: A unilateral cerebellar montage with the anode three cm lateral to the inion on the side ipsilateral to the more PD-affected side and the cathode on the ipsilateral cheek. Stimulation is ramped up to 4 mA over the first 30 seconds and stays at 4 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 4 mA: Uses weak electrical current (4 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
- Bilateral, 4 mA: Bilateral cerebellar tDCS will have both electrodes placed 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is ramped up to 4 mA over the first 30 seconds and stays at 4 mA for the remainder of the stimulation time.
  Transcranial direct current stimulation at 4 mA: Uses weak electrical current (4 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
Arm/Group | Sham | Unilateral, 2 mA | Bilateral, 2 mA | Unilateral, 4 mA | Bilateral, 4 mA
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT04046055/Prot_SAP_001.pdf